CLINICAL TRIAL: NCT04193423
Title: Deep Cervical Flexors or Cervical Extensors Strengthening Program in Patients With Chronic Neck Pain, Does it Matter Which One to Choose?: A Randomized Clinical Trial
Brief Title: The Effects of Exercise Therapy for Flexor and Extensor Cervical Muscles on Non-specific Neck Pain.
Acronym: CCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/28; U1111-1241-3966 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain; Chronic Pain
Keywords: neck pain; exercise; training; endurance; intervention
MeSH Terms: conditions — Neck Pain; Chronic Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled clinical trial with parallel groups.
Who Masked: Participant
Masking Description: It is a single-blind study: only the investigator performing the measurements will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A-Group: craniocervical and cervicothoracic extension training (Experimental)
  Interventions: Other: Neck extensors training versus deep cervical flexors training, compared to a control group.
- B-Group: craniocervical flexion training (Experimental)
  Interventions: Other: Neck extensors training versus deep cervical flexors training, compared to a control group.
- C-Group: control group (Active Comparator): No intervention will be performed due to the fact that they will be still on the waiting list.
  Interventions: Other: Neck extensors training versus deep cervical flexors training, compared to a control group.

INTERVENTIONS:
Other: Neck extensors training versus deep cervical flexors training, compared to a control group. — During the first month, the participants of the experimental groups will come at Rehabilitation Service to do the exercises individually and supervised by the physiotherapist and to received the conventional treatment (10 minutes of infrared heat, 10 minutes of massage and 15 minutes of TENS). The last six months, they will perform daily home exercises.
  * A-group: the degrees respect to the floor in wich each participant can hold the craniocervical extension and the cervicothoracic extension during 5 seconds will bo measured with the BDI.
  * B-group: Using an air-filled pressure sensor placed behind the neck, the physiotherapist will identify the target level that the patient can hold steadily a craniocervical flexion (CCF) for 5 seconds in a controlled manner. They will train following the protocol described by Jull et al.
  Of each of this exercises, they will perform 10 isometric contractions, at the corresponding degrees or target level, of 10 seconds with a rest of 3-5 seconds.

SUMMARY:
Objective:

To compare the effects craniocervical and cervicothoracic extension training versus deep cervical flexor training, both combined with conventional treatment, on disability, perceived pain, Health-related quality of life (HRQoL), endurance, active range of motion (AROM) of the cervical spine, joint position sense (JPS) and intake of drugs in subjects with non-specific chronic neck pain, referenced by the control group.

Methods:

The research will be done from December 2019 to August 2020 at the Recoletas Burgos Hospital.

Fifty-four volunteers with non-specific chronic neck pain, recruited at the hospital, will be randomly assigned, using sealed envelopes, to 1 of the three groups.

The first two experimental groups will be named Group A and Group B and each of them will go to the Rehabilitation Service for 4 weeks to perform the exercises under the supervision of the physiotherapist. This process will occur along with the conventional treatment (infrared heat, massage and transcutaneous electrical nerve stimulation). These groups will differ between them in the muscles they will mainly train through training. The group A will perform a neck extensor muscles training and group B a deep cervical flexor muscles training. After these 4 weeks, these exercises will be performed by them on a daily routine which will be prescribed for 6 months at home.

On the control group (group C), no intervention will be performed due to the fact that they will be still on the waiting list.

Disability, pain, HRQoL and drug intake will be measured in pre-treatment, at 4 weeks (post-treatment) and at 6 months follow-up; endurance, AROM and JPS will be measured in pre-treatment and at 4 weeks (post-treatment); while demographic variables (height, weight and age) will only be measured at the baseline.

ELIGIBILITY:
Inclusion Criteria:

* non-specific neck pain (NSNP) for at least 3 months prior intervention commencement,
* age between 18 and 65 years,
* sedentary lifestyle,
* score > 5/50 on the Neck Disability Index (NDI) or score > 2 on the Numeric Rating Scale (NPRS) whose symptoms are not increased performing the exercises proposed in the study,
* limitation in the Active Range of cervical Motion (AROM) in flexion, extension, lateral inclination and/or rotation.

Exclusion Criteria:

* previous neck surgery,
* neck pain associated with whiplash injuries,
* subjects who ave received physical therapy 3 months prior intervention commencement,
* dizziness in the quadruped position, supine position, sitting or performing neck movements,
* pain in other parts od the body that prevents the performance of the exercises proposed in the study,
* neck pain accompanied by vertigo caused by vertebrobasilar insufficiency or pain accompanied by non-cervicogenic headaches,
* neck pain with cervical radiculopathy and/or externalized cervical disc herniation,
* red flags: fracture, tumor or cervical infection or diagnosis of osteoporosis, metabolic diseases or rheumatoid arthritis,
* myopathy, ankylosing spondylitis or fibromyalgia,
* central nervous system involvement,
* pregnant women,
* severe psychiatric oe psychological disorders,
* subjects with pending legal action,
* not understand, write and speak spanish fluently.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Change in Pain related disability | Baseline, 1 month (primary timepoint) and 6 months after intervention.
  using the Neck Disability Index (NDI) Questionnaire

SECONDARY OUTCOMES:
Change in Neck pain | Baseline, 1 month (primary timepoint) and 6 months after intervention.
  Using a Numeric Rating Scale (NPRS) from 0 to 10
Change in Health-related quality of life (HRQoL) | Baseline, 1 month (primary timepoint) and 6 months after intervention.
  using the SF-36 quality of life questionnaire.
Change in Neck muscles endurance | Baseline and 1 month (primary timepoint).
  Using the modified Neck Extensor Endurance test (NEE test) proposed by Lee el al. (2005) or the Neck Flexor Muscle Endurance Test (NFME test) with a chronometer and a BDI
Change in Active Range of cervical Motion (AROM) | Baseline and 1 month (primary timepoint).
  Using a digital inclinometer
Change in Joint Position Sense (JPS) | Baseline and 1 month (primary timepoint).
  Using a target and a rule
Change in Frequency of use of drugs | Baseline, 1 month (primary timepoint) and 6 months after intervention.
  Using a shelf-completed drug registration document

CONTACTS AND LOCATIONS:
Overall Officials: Achalandabaso, Study Director — University of Jaén
Locations (1):
- Recoletas Burgos Hospital, Burgos, Spain